CLINICAL TRIAL: NCT06162039
Title: Prevalence of Hemorrhagic Myocardial Infarction in the United States
Brief Title: National Landscape of Hemorrhagic Myocardial Infarction in the United States
Acronym: MIRON-NATIONAL
Status: Completed | Type: Observational
Sponsor: Rohan Dharmakumar (Other)
Responsible Party: Sponsor-Investigator, Rohan Dharmakumar, Executive Director, Medical Imaging Research Institute, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: 19978b
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Registry analysis for prevalence of hemorrhagic myocardial infarction in the United States

ELIGIBILITY:
Inclusion Criteria:

* Acute Myocardial Infarction - STEMI Primary PCI Availability of lab parameters and/or CMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All STEMI who underwent primary coronary intervention and revascularisation
Sampling Method: Non-Probability Sample
Enrollment: 24181 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Statewise proportion of Hemorrhagic Myocardial Infarction in the United States | 10 years
  Prevalence of Hemorrhagic Myocardial Infarction

SECONDARY OUTCOMES:
Statewise proportion of Acute Heart Failure in Hemorrhagic Myocardial Infarction | 30 days
  Prevalence of Acute Heart Failure in Hemorrhagic Myocardial Infarction
Statewise proportion of re-hospitalization in Hemorrhagic Myocardial Infarction | 30 days
  Prevalence of re-hospitalization in Hemorrhagic Myocardial Infarction
Statewise proportion of arrhythmia in Hemorrhagic Myocardial Infarction | 30 days
  Prevalence of arrhythmia in Hemorrhagic Myocardial Infarction

CONTACTS AND LOCATIONS:
Overall Officials: Keyur P Vora, MD FACC, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Medical Imaging Research Institute, Cardiovascular Imaging Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No